CLINICAL TRIAL: NCT05451342
Title: Explore Potential Plasma and BALF Immunometabolic and Lipidomic Biomarkers for Identifying the Endotypes in Patients With ARDS
Brief Title: Explore Potential Plasma and BALF Immunometabolic and Lipidomic Biomarkers for Identifying ARDS Endotypes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZS-3391
Record Dates: First submitted 2022-06-27; First posted 2022-07-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-06

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Respiratory Failure
Keywords: ARDS, biomarkers, immunometabolism
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARDS: Patients who meet the diagnostic criteria of ARDS
  Interventions: Diagnostic Test: Integrated Transcriptomics, Metabolomics, and Lipidomics Profiling
- Non-ARDS: Patients without ARDS
  Interventions: Diagnostic Test: Integrated Transcriptomics, Metabolomics, and Lipidomics Profiling

INTERVENTIONS:
Diagnostic Test: Integrated Transcriptomics, Metabolomics, and Lipidomics Profiling — Blood samples and BALD samples will be collected for further integrated transcriptomics, metabolomics, lipidomics analysis, and exosome extraction.

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a life-threatening condition that causes high mortality (41% to 58%). Previous studies have reported that biomarkers can facilitate phenotypic diagnosis of ARDS, enabling precision treatment of ARDS. Although there were many studies that found some potential therapeutic targets for ARDS, no pharmacotherapies have been validated to treat ARDS. The development of biomarkers to predict the prognosis and monitor the response to treatment would be of interest for selecting patients for specific therapeutic trials. Many recent studies have shown that immune metabolic changes are involved in the pathogenesis of ARDS and may become a new therapeutic target for them. We aimed to identify a panel of immunometabolic and lipidomic biomarkers derived from blood and bronchoalveolar lavage fluid (BALF) which may help differentiate the ARDS endotypes.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is an observational study. The blood and BALF samples will be collected from patients with ARDS for exosome extraction and transcriptome and metabolomic analysis.

Exosome characterization and differential genes and metabolites will be identified.

ELIGIBILITY:
Inclusion Criteria:

1. Aged >18 years old;
2. Meet the diagnostic criteria of ARDS according to the Berlin Criteria.

Exclusion Criteria:

1. Aged≤18 years old;
2. Pregnancy;
3. No informed consent;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients with the diagnosis of ARDS
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Identification of ARDS Endotypes | 2 years
  Blood samples will be collected on day 1, 3, 5,7 since ARDS diagnosis is made (day 0) and BALF samples will be collected on day 1 and day 7. Blood samples are used to extract PBMC and BALF samples are used to extract alveolar macrophage. Afterwards, PBMC and alveolar macrophage are saved for further transcriptomic and metabomic analysis. At the same time, clinical and biological date are collected to identify subgroups of patients that might share mortality risk, clinical course, and/or treatment responsiveness. At last, the relationship between transcriptomic and metabomic signature of PBMC and alveolar macrophage and the clinical phenotypes are analyzed to determine ARDS endotypes.

SECONDARY OUTCOMES:
Compare the PBMC and alveolar macrophage derived exosome levels between patients with ARDS and without ARDS | 2 years
  Plasma and BLAF supernatant are used for exosome extraction
Correlation of Endotypes with published ARDS specific Biomarkers | 2 years
  Correlate the endotypes with published markers of hyperinflammatory, microvascular-injury predominant, and distal lung epithelial cell-predominant injury in ARDS
Correlation of Endotypes with Intensive care unit-free days | Until 28 days following ICU admission
  Intensive care unit-free days are calculated by the number of days in the first 28 days following ICU admission that a patient is alive and not in the intensive care unit.
Correlation of Endotypes with Ventilator-free days | Until 28 days following ICU admission
  Ventilator-free days are calculated by the number of days in the first 28 days following ICU admissionthat a patient is alive and not on a ventilator.
Correlation of Endotypes with All-cause mortality | Until death or hospital discharge, assessed up to 28 days following ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, MD, Study Director — Peking Union Medical College
Locations (2):
- China (2):
  - PUMC, Beijing, Beijing Municipality
  - Yingying Yang, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No